CLINICAL TRIAL: NCT03426813
Title: Is There an Effect of Early Mobilization of Patients With Community-acquired Pneumonia?
Brief Title: Early Mobilization of Patients With Community-acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Dorte Melgaard Kristiansen, Development therapist, Regionshospital Nordjylland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHN_DMK_04
Record Dates: First submitted 2012-12-20; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Pneumonia
Keywords: mobilization; physiotherapy; community-acquired pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early mobilization (Other): Historical control group for early mobilization
  Interventions: Other: Historical control group for early mobilization

INTERVENTIONS:
Other: Historical control group for early mobilization

SUMMARY:
Pneumonia is a common health problem.This thesis may clarify whether early mobilization influence the time these patients are hospitalized, whether they are rehospitalized and whether it is possible to reduce the mortality rate.

DETAILED DESCRIPTION:
Pneumonia is a common health problem. More than 100,000 Danes contract pneumonia every year, and around 15,000 of these are hospitalized. The main treatment is antibiotics. An American study indicates that patients who are mobilized early are hospitalized for a shorter period of time. The objective of the thesis is: to determine the effect of mobilization within 24 hours after hospitalization of patients with pneumonia. The result will be number of hospitalization days, rehospitalisation and mortality.

Patients with pneumonia hospitalized in the period 1 September 2012 - 28 February 2013 in the Medical Centre, lung unit 204B at Vendsyssel Hospital will be included in the project. Within the first 24 hours of hospitalization, they will be tested by a physiotherapist and mobilized.

There are significant costs associated with the treatment of patients with pneumonia - both economic costs and human costs. This thesis may clarify whether early mobilization influence the time these patients are hospitalized, whether they are rehospitalized and whether it is possible to reduce the mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* patients with community-acquired pneumonia

Exclusion Criteria:

* dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The number of hospitalization days | 6 months
  Length of stay

SECONDARY OUTCOMES:
Number of rehospitalizations | 6 months after 1st hospitalization
  Rehospitalizations

OTHER OUTCOMES:
Mortality | 6 months after 1st hospitalization
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- North Denmark Hospital, Hjørring, Denmark